CLINICAL TRIAL: NCT06699199
Title: Effect of Silver Diamine Fluoride Application on Oral Microbiome of Saudi Children: Randomized Clinical Trial in Jeddah City
Brief Title: Effect of Silver Diamine Fluoride Application on Oral Microbiome of Healthy Pediatric Patient
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Collaborators: King Fahd Medical Research Centre (Other)
Responsible Party: Principal Investigator, Doaa Yasir Jamal, PhD candidate - Pediatric dental specialist, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 139-07-23; Research center (Other: King fahad medical research center, Dr. Turki Abujamel)
Record Dates: First submitted 2024-11-09; First posted 2024-11-21 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-11

CONDITIONS: Dental Caries
Keywords: Dental Management; Oral Microbiome; Caries Arrest; SDF; Silver diamine fluoride 38%; Potassium iodide
MeSH Terms: conditions — Dental Caries | interventions — silver diamine fluoride; Potassium Iodide

STUDY DESIGN:
Intervention Model Description: Children will receive one of two interventions
  1. Silver diamine fluoride 38% (SDF only) or,
  2. Silver diamine fluoride 38% + potassium iodide (SDF +KI) Both treatment are recommend and approved as an arresting treatment of Dental caries in children as an intermediate management
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arresting Treatment 1 (Active Comparator): Management of dental caries in children between the ages of 4 and 10 by arresting the lesion using standard Treatment for caries arrest, which is silver diamine fluoride %38
  Interventions: Drug: Silver diamine Fluoride 38%
- Arresting Treatment 2 (Experimental): Management of dental caries n children between the ages of 4 and 10 by arresting the lesion using an alternative Treatment by using the combination of Silver diamine fluoride 38% + potassium iodide (SDF+KI), Both products reported as materials with an anti-microbial effect
  Interventions: Drug: Silver diamine fluoride- potassium iodide

INTERVENTIONS:
Drug: Silver diamine Fluoride 38% — Intervention is the application of Silver diamine fluoride 38% to children Group in arm 1 (Arm 1): children will receive Silver diamine fluoride 38% application for 1 min to arrest primary teeth
  SDF: (Silver diamine fluoride 38% is a material used for arresting caries lesions in primary and permanent teeth)
  - SDF Product generic name and information (E-SDF: it is a 1-step Technique) - The 38% SDF solution comprised a blend of silver, fluoride, and ammonia at a total concentration of 38%.
  Other Names: E-SDF; Silver diamine fluoride
  Arms: Arresting Treatment 1
Drug: Silver diamine fluoride- potassium iodide — Intervention is the application of Silver diamine fluoride 38% + potassium iodide to children Group in arm 2 (Arm 2): children will receive Silver diamine fluoride 38% application for 1 min to arrest primary teeth, Followed by an second minute of potassium iodide solution application
  - SDF Product generic name and information (Riva-star: it is a 2-step Technique) 30-35% SDF solution (1st step) comprised a blend of silver, fluoride, and ammonia applied in combination with a second application of potassium iodide solution (2nd step)
  Other Names: Silver diamine fluoride 38% + potassium iodide; Riva- star SDF
  Arms: Arresting Treatment 2

SUMMARY:
This clinical trial aims to learn more about the working mechanism of an antimicrobial agent used to manage dental caries, especially in young, uncooperative children. It will also provide a deeper insight into different products of the same agent and its effectiveness in Arresting dental caries.

The main questions it aims to answer are:

What is the clinical impact of silver diamine fluoride application in caries-active children? What is the antimicrobial effect of silver diamine fluoride in oral microbial inhabitants? Researchers will compare silver diamine fluoride (SDF)only and silver diamine fluoride+ potassium iodide(SDF+KI) to see which materials substantially affect on dental caries and oral microbial inhabitants

Participants/Parent will:

The parent will fill out a comprehensive data sheet for the child (childhood and current dental and medical history) Visit the dental clinic to Receive one of 2 (SDF or SDF+KI) treatment applications once Visit the clinic a 2nd time for a 2-4 week Treatment Follow-up Go through the sample collection process twice( pre- and 2-4 weeks post- Treatment) Sample collection including (Saliva- Biofilm and caries tissue sample)

DETAILED DESCRIPTION:
Aim of the Work

This study aims to:

1. Evaluate the Arresting effect of 1-step (SDF only) versus 2-step (SDF+KI) application.
2. Explore the effectiveness of SDF compared to SDF+KI on oral Microbiome.
3. Evaluate and compare saliva composition before and after SDF application. Study Question What is the clinical and laboratory impact of silver diamine fluoride application in caries-active children? Research Null Hypothesis

<!-- -->

1. There is no difference in the Arresting effect of SDF versus SDF+KI application.
2. There is no difference between the effectiveness of SDF versus SDF+KI application on oral Microbiome.
3. There is no difference in in saliva composition before and after SDF

Research protocol:

Materials and methods The study will be conducted at the Department of Pediatric Dentistry, Faculty of Dentistry, King Abdul Aziz University, after approval from the University Institutional Ethics Committee.Informed consent will be obtained from the participant's parent. The sample will be collected, and sent to King Fahd Medical Research Center

Patients' enrollment An informed consent document will be obtained from those participant parents willing to be part of the trial before the study start. A brief interview-based survey will be conducted about general and dental health, oral hygiene, sugar consumption, and family demographics. A calibrated pediatric dentist will do dental examinations and lesion evaluations, followed by sample collection.

Biospecimens collection protocol:

* All participants will be required to fast for 90 minutes prior to specimen collection.
* All participants will be seated in an upright position in the dental chair.
* Sample will be collected in the first visit for all children, and another set of samples will be collected again for children recruited in the second part of the study.
* Each child will have an oral swab, saliva, supragingival plaque, and subsurface dentine obtained. The collection will be conducted in the following manner:

  1. Saliva sample ▪ Unstimulated saliva (S, Saliva) will be obtained from enrolled children. using a standardized Spitting method

     ▪ Approximately 5 ml of un-stimulated saliva will be collected using 50 ml falcon tube/ specimen container.

     ▪ Collected saliva will transferred and stored in an Eppendorf tube using 5-10 ml syringe.
  2. Biofilm samples

     ▪ Biofilm samples will be collected from both teeth with and without Carious surfaces.

     ▪ Sterilized Microbrush/paper points will be used for collection of dental plaque
  3. Subsurface carious dentin ▪ Sample collection from within the extensive untreated caries (at baseline visit) ▪ Sterilized dental excavators and sterilized large round bur will be used for sample collection▪ Subsurface carious dentin excavation utilizing a spoon excavator and round bur to extract carious dentin tissue (1.0 to 1.5 mm of depth) Collection and storage procedure The sample will be collected from recruited children at the first visit (as the baseline).

A sterilized dental instrument will be used for the collection of samples, The samples will be stored in Eppendorf tubes filled with 200LμL of phosphate-buffered saline (PBS) solution. Before laboratory analysis, all gathered samples will be kept in a freezer at - 80 °C.

Clinical trial PICO:

P: Children aged 2-10 years caries-free or with caries- active (with at least 1 tooth with deep cavitated lesions (with no signs of pulpitis)) I: Management using SDF (Silver diamine fluoride 38%) C: Management using a different fluoride containing product (SDF 38%+KI) O: Alteration in metabolomics and microbiome.

Patients' enrollment At the first visit, children with active dental caries will undergo a sample collection process conducted by a calibrated pediatric dentist who will also provide the intervention treatment during the same session (baseline visit). A second sample collection appointment will be scheduled after two to three weeks, followed by another follow up visit after two-week.

Study groups:

* Experiment group The intervention participant will receive silver diamine fluoride 38%
* Comparison group The Comparison participant will receive SDF+KI system. Intervention A calibrated pediatric dentist will perform the procedures. Saliva and plaque sample will be collected on completion of SDF application.

Sample collection:

* Sample collection will be conducted Before, 2 and 4 weeks after Intervention.
* The sample included are saliva, supragingival and occlusal plaque, caries plaque (Carious and SDF-treated surfaces), and subsurface carious dentin (from within the carious untreated lesion)▪ Plaque Sample of supragingival and occlusal plaque will be collected from primary and permanent teeth. Outcomes The primary outcome measure will be the difference in microbiome groups over time and the difference within the treatment groups. The secondary outcome will be the effect on salivary metabolomics.

Assessment will include:

1. The microbial community composition of surface biofilm prior to and post SDF treatment.

2. Subsurface microbiota and microbial community composition prior and post SDF treatment.

3. Comparing the microbial community composition of dentin&#39;s subsurface microbiota after treatment with SDF and SDF+KI. 4. Salivary metabolomics before and after SDF Statistical Analyses Continuous data will be reported as means and standard deviations, whereas categorical variables will be presented as frequencies and percentages (SD). Statistical significance across groups will be determined using either a one-way analysis of variance (ANOVA) model or the non-parametric version of the Kruskal-Wallis test, depending on whether the variables are normally distributed. Using R, taxonomy plots and tables will be generated, and relative abundance at different taxonomic levels and microbial diversity indices will be calculated. Between the groups, relative abundance and alpha and beta diversity parameters will be evaluated. In addition, the relationship between caries activity, caries risk factors, clinical features, and microbiota composition will be studied prior to and following intervention. Statistical significance will be regarded when p-values are less than 0.05, and P-values in multiple comparisons will be adjusted for the false discovery rate (FDR). Expected Findings:1. There is a difference in the clinical and microbial effect of SDF versus SDF+KI application on oral microbiome 2. There is a shift in saliva composition before and after SDF.

ELIGIBILITY:
Inclusion criteria

* Healthy patients.
* Patients within 4-10 years of age.
* The presence of at least one deciduous tooth with a caries lesion that is directly accessible (cavitates)

Exclusion Criteria:

* Presentation of irreversible pulpititis or necrosis• The extensive lesion was restored.
* The surface of the lesion was hard and smooth.
* Children with inherited or systemic conditions.
* Children with a substantial medication history or those who have taken antibiotics within the previous three months.
* Children who have undergone topical fluoride treatment within the previous 2 weeks.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Arresting Effect | Baseline and follow up (after 2-4 weeks)
  Arresting conditions (Arresting rate) will be assessed through clinical examination and intra-oral Photos evaluation of the cavities before and 2-4 weeks after SDF treatments
  * Caries activity status will be recorded as (active;1 or arrested;2) according to hardness and color (Caries activity status scored as 1: active or 2: arrested
  * Descriptive definition :
    * 1:Active lesion: tooth surface is deemed active if any softened area on the carious lesion is detected upon probing or no obvious changes in color, and the lesion is still soft.
    * 2:Arrested lesion: When the entire carious lesion is determined to be hard upon probing, or lesion is Darker in color and has hard surfaces (harder to excavate with a spoon excavator), it will be recorded as arrested caries.

SECONDARY OUTCOMES:
Microbial status | Baseline and follow up (after 2-4 weeks)
  Change in oral Microbial inhabits using sequencing techniques of the oral Microbiome. Microbial DNA will be extracted and sequenced using 16S rRNA gene amplicon-based and shotgun metagenomic sequences.
  Data will be presented as
  1. Changes of microbial taxonomic profiles and microbial diversity within the same group (SDF group or SDF+KI group)
  2. Difference in microbial taxonomic profiles and microbial diversity between interventions groups after assigned treatment application, differences between groups (SDF group and SDF+KI group)

OTHER OUTCOMES:
Adverse events | Baseline and follow up (after 2-4 weeks)
  Any reported outcome by the child or parents of the following; (by answering a yes or no questions in a follow up visit short interview based questionnaire)
  * Pain/ sensitivity: (Yes or No)
  * Discoloration/stains other areas (Extra- Intra):(Yes or No)
  * Metallic taste: (Yes or No)
  * Gingival lesions: (Yes or No)
  * Pulp or abscess: (Yes or No)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Turki S Abujamel, BDS, MSc, PhD, Study Director — Department of Medical Laboratory Science, King Abdulaziz University and KFMRC Deputy Director of Administrative and Financial Affairs.; Prof. (Dr.) Abdullah S AlMushayt, BDS, MSc, PhD, Study Director — Faculty of Dentistry, Department of Pediatric Dentistry, King Abdulaziz University Jeddah, Saudi Arabia; Nada O Bamashmous, BDS, MSc, DDENT, Study Director — Faculty of Dentistry, Department of Pediatric Dentistry, King Abdulaziz University Jeddah, Saudi Arabia; Shatha O Bamashmous, BDS, MSc, PhD, Study Director — Department of Periodontology, KAU Faculty of Dentistry, Jeddah, Saudi Arabia
Locations (1):
- University Dental hospital of King Abdulaziz University, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
The quantity of patient data to be provided has not yet been determined. Prior to confirming any plans for sharing patient information, the Organisation will thoroughly assess and approve the data sharing process to guarantee compliance with patient confidentiality rights.